CLINICAL TRIAL: NCT01778114
Title: Bioavailability of Vitamin D2 and Vitamin D3 in Supplements Compared to Vitamin D3 and Vitamin D2 in Fortified Orange Juice
Brief Title: Availability of Vitamin D in Orange Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Michael F. Holick, Michael . Holick PhD, MD, Boston University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H-26117
Record Dates: First submitted 2013-01-23; First posted 2013-01-29 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D2; Vitamin D3; Vitamin D; Orange Juice
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo + orange juice without vitamin D (Placebo Comparator): Placebo + orange juice without vitamin D
  Interventions: Other: Placebo
- Placebo + 1000 IU vitamin D3 in OJ (Experimental): Vitamin D3 in orange juice
  Interventions: Dietary Supplement: Vitamin D3 in orange juice
- Placebo + 1000 IU vitamin D2 in OJ (Experimental): Vitamin D2 in orange juice
  Interventions: Dietary Supplement: Vitamin D2 in orange juice
- 1000 IU vitamin D3 + placebo OJ (Active Comparator): 1000 IU vitamin D3 + placebo OJ
  Interventions: Dietary Supplement: Vitamin D3
- 1000 IU vitamin D2 + placebo OJ (Active Comparator): 1000 IU vitamin D2 + placebo OJ
  Interventions: Dietary Supplement: Vitamin D2

INTERVENTIONS:
Dietary Supplement: Vitamin D2 in orange juice — 1000 IU dose
  Arms: Placebo + 1000 IU vitamin D2 in OJ
Dietary Supplement: Vitamin D3 in orange juice — 1000 IU
  Arms: Placebo + 1000 IU vitamin D3 in OJ
Dietary Supplement: Vitamin D2 — capsule, 1000 IU
  Arms: 1000 IU vitamin D2 + placebo OJ
Dietary Supplement: Vitamin D3 — capsule, 1000 IU
  Arms: 1000 IU vitamin D3 + placebo OJ
Other: Placebo — Placebo
  Arms: Placebo + orange juice without vitamin D

SUMMARY:
The purpose of this study was to determine whether vitamin D2 and vitamin D3 in orange juice are effective at raising vitamin D levels in the blood and if vitamin D2 and vitamin D3 in orange juice raised blood levels of 25(OH)D as well as vitamin D3 and vitamin D2 supplements.

DETAILED DESCRIPTION:
This study should provide valuable information about the bioavailability of both vitamin D2 and vitamin D3 formulated in orange juice compared to vitamin D2 and vitamin D3 formulated in a pill and taken with water. It is anticipated based on our previous observation that the vitamin D2 and vitamin D3 in orange juice will be at least 50% more effective in raising the blood levels of 25(OH)D than when taken in pill form.

This study will evaluate the bioavailability and metabolism of vitamin D2 and vitamin D3 in combination in tablet form. The results should provide important information as to whether a physiologic dose of vitamin D2 has a negative effect on circulating levels of 25-hydroxyvitamin D2 [25(OH)D2 ] and on 25-hydroxyvitamin D3 [25(OH)D3]. Results from this study have important implications for expanding the adequate intake (AI) recommendations for vitamin D2 and vitamin D3 for adults.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults of all races ages 18 years and older

Exclusion Criteria:

* Pregnant and lactating women
* History of chronic severe liver (as defined by liver function test greater than 2 times upper limit of normal)or kidney disease as defined by a serum creatinine >2.5.
* History of taking a daily supplement that contains 400 or more IU vitamin D2 or vitamin D3 within the past month or taking a pharmacologic amount of vitamin D2 or one of the active vitamin D analogs including Zemplar (Paricalcitol), Dovonex (calcipotriol), Hectorol (vitamin D pro hormone)
* Subjects who are taking orally Dilantin or glucocorticoids.
* Exposure to a tanning bed or tanning on a beach for more than eight hours within the past month.
* Subjects who drink more than 2 glasses (16 oz) cups of milk a day.
* Known history of elevated calcium. (> 10.5 mg% (mg/dl))
* History of intestinal malabsorption (i.e. Cystic Fibrosis, Fat malabsorption Syndrome, Crohn's Disease)
* Allergies to orange juice
* Any medical conditions in which it is not advisable to receive one 8 oz. glass of orange juice per day.
* Currently taking, or having taken less than one month prior to start of study, a prescription vitamin D
* Unwilling to consent to this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-12; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Measurement of 25(OH)D levels after ingestion of 1,000 IU of vitamin D2 or vitamin D3 in a capsule | 11 weeks

SECONDARY OUTCOMES:
Measurement 25(OH)D levels after taking vitamin D2 or vitamin D3 in orange juice | 11 weeks

OTHER OUTCOMES:
Compare 25(OH)D levels in subjects taking vitamin D2 versus vitamin D3 | 11 weeks
  It is debated in the literature that vitamin D2 is more effective than vitamin D3 in maintaining 25(OH)D levels in the blood. This outcome measure will help determine if this is true or if they are equally effective.
Determine serum 1,25(OH)2D levels | 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, PhD, MD, Principal Investigator — Boston University; Rachael M Biancuzzo, BS, MA, Study Director — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holick MF. High prevalence of vitamin D inadequacy and implications for health. Mayo Clin Proc. 2006 Mar;81(3):353-73. doi: 10.4065/81.3.353. PMID 16529140
- [Background] Holick MF. Sunlight "D"ilemma: risk of skin cancer or bone disease and muscle weakness. Lancet. 2001 Jan 6;357(9249):4-6. doi: 10.1016/S0140-6736(00)03560-1. No abstract available. PMID 11197362
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes. Dietary Reference Intakes for Calcium, Phosphorus, Magnesium, Vitamin D, and Fluoride. Washington (DC): National Academies Press (US); 1997. Available from http://www.ncbi.nlm.nih.gov/books/NBK109825/ PMID 23115811
- [Background] Webb AR, Kline L, Holick MF. Influence of season and latitude on the cutaneous synthesis of vitamin D3: exposure to winter sunlight in Boston and Edmonton will not promote vitamin D3 synthesis in human skin. J Clin Endocrinol Metab. 1988 Aug;67(2):373-8. doi: 10.1210/jcem-67-2-373. PMID 2839537
- [Background] Malabanan A, Veronikis IE, Holick MF. Redefining vitamin D insufficiency. Lancet. 1998 Mar 14;351(9105):805-6. doi: 10.1016/s0140-6736(05)78933-9. No abstract available. PMID 9519960
- [Background] Tangpricha V, Koutkia P, Rieke SM, Chen TC, Perez AA, Holick MF. Fortification of orange juice with vitamin D: a novel approach for enhancing vitamin D nutritional health. Am J Clin Nutr. 2003 Jun;77(6):1478-83. doi: 10.1093/ajcn/77.6.1478. PMID 12791627
- [Background] Holick MF, Siris ES, Binkley N, Beard MK, Khan A, Katzer JT, Petruschke RA, Chen E, de Papp AE. Prevalence of Vitamin D inadequacy among postmenopausal North American women receiving osteoporosis therapy. J Clin Endocrinol Metab. 2005 Jun;90(6):3215-24. doi: 10.1210/jc.2004-2364. Epub 2005 Mar 29. PMID 15797954
- [Background] Heaney RP, Davies KM, Chen TC, Holick MF, Barger-Lux MJ. Human serum 25-hydroxycholecalciferol response to extended oral dosing with cholecalciferol. Am J Clin Nutr. 2003 Jan;77(1):204-10. doi: 10.1093/ajcn/77.1.204. PMID 12499343
- [Background] Armas LA, Hollis BW, Heaney RP. Vitamin D2 is much less effective than vitamin D3 in humans. J Clin Endocrinol Metab. 2004 Nov;89(11):5387-91. doi: 10.1210/jc.2004-0360. PMID 15531486
- [Background] Trang HM, Cole DE, Rubin LA, Pierratos A, Siu S, Vieth R. Evidence that vitamin D3 increases serum 25-hydroxyvitamin D more efficiently than does vitamin D2. Am J Clin Nutr. 1998 Oct;68(4):854-8. doi: 10.1093/ajcn/68.4.854. PMID 9771862
- [Result] Biancuzzo RM, Young A, Bibuld D, Cai MH, Winter MR, Klein EK, Ameri A, Reitz R, Salameh W, Chen TC, Holick MF. Fortification of orange juice with vitamin D(2) or vitamin D(3) is as effective as an oral supplement in maintaining vitamin D status in adults. Am J Clin Nutr. 2010 Jun;91(6):1621-6. doi: 10.3945/ajcn.2009.27972. Epub 2010 Apr 28. PMID 20427729